CLINICAL TRIAL: NCT06167707
Title: Open-label, Single-dose, Randomized, Two-way Crossover Study to Compare the Pharmacokinetics and Pharmacodynamics of Subcutaneous Injection of SCP-111 (Furosemide) vs Intravenous Injection of Furosemide in Healthy Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics of Subcutaneous vs Intravenous Furosemide in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: scPharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: scP-04-001
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure; Fluid Overload
MeSH Terms: conditions — Heart Failure; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1 (Experimental): Period 1: SC Period 2: IV
  Interventions: Drug: SCP-111; Drug: Furosemide USP
- Treatment Sequence 2 (Experimental): Period 1: IV Period 2: SC
  Interventions: Drug: SCP-111; Drug: Furosemide USP

INTERVENTIONS:
Drug: SCP-111 — Furosemide injection 80 mg/mL, 80 mg SC via autoinjector x 1 dose
Drug: Furosemide USP — Furosemide injection, USP 10 mg/mL, 40 mg IV over 2 minutes followed by 40 mg 2 hours later

SUMMARY:
This study aims to compare the pharmacokinetics and pharmacodynamics of intravenous (IV) and subcutaneous (SC) furosemide. The test formulation in this study is furosemide injection, 80 mg/1 mL, buffered to a neutral pH for SC administration via an autoinjector. A commercial formulation of furosemide injection, USP, solution 10 mg/mL administered as a 40 mg IV injection over 2 minutes followed by a second dose of 40 mg, 2 hours later, will serve as the reference drug.

The objectives of this study are:

* To estimate the bioavailability and describe the pharmacokinetics and pharmacodynamics of furosemide administered as SC injection via autoinjector compared with equivalent dose of furosemide administered as two 40 mg IV injections, two hours apart.
* To describe the safety and tolerability of furosemide administered as SC injection via an autoinjector.

DETAILED DESCRIPTION:
This is an open-label, single-center, single-dose, randomized, two-way crossover study in healthy volunteers. Each Subject will complete Screening, Baseline, Treatment, and Follow-up Phases.

After a Screening Phase, Subjects meeting entry criteria will be admitted to the clinical research unit (CRU) and undergo baseline assessments. Subjects will be randomly assigned in a 1:1 ratio to 1 of 2 treatment sequences (IV furosemide followed by SC or vice versa). Subjects will remain domiciled in the CRU for each treatment period which will be about 12-hours. After final assessments are performed, Subjects may be discharged from the CRU if safety parameters are acceptable to the Investigator and return to the CRU after a 3-day washout period to receive the second treatment sequence. The Follow-up Phase will occur 24-48 hours after discharge from the CRU following treatment sequence 2, completing Subjects' study participation.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
2. Male and female subjects 45 to 80 years of age.
3. Has the ability to understand the requirements of the study and is willing to comply with all study procedures.
4. In the opinion of the Investigator, able to participate in the study.

Exclusion Criteria:

1. Pregnant or lactating women or women of childbearing age who are not willing to use an adequate form of contraception.
2. Systolic BP (SBP) < 90 mmHg at screening or baseline.
3. Heart rate > 110 beats per minute (BPM) at screening or baseline.
4. Temperature > 38°C (oral or equivalent).
5. Serum potassium < 3.0 or > 5.5 mEq/L at screening.
6. Other significant cardiac abnormalities which may interfere with study participation or study assessments.
7. Current or planned treatment during the study with any IV therapies, including inotropic agents, vasopressors, levosimendan, nesiritide or analogues. scPharmaceuticals, Inc. SCP-111 PK/PD Study Protocol Number: scP-04-001 Confidential Page 14 of 56
8. Presence of implanted ventricular assist device, cardiac defibrillator or pacemaker.
9. Severely impaired renal function, defined as an estimated glomerular filtration rate (eGFR) at screening admission < 30 mL/min/1.73m2, calculated using the simplified Modification of Diet in Renal Disease (sMDRD) equation.
10. Urinary retention due to bladder emptying disorders and/or urethral narrowing.
11. Presence or need for urinary catheterization.
12. Reported history of hepatic cirrhosis.
13. Administration of intravenous radiographic contrast agent within 72 hours prior to Screening.
14. Concomitant or any use within past 30 days of drugs known to interact with furosemide (aminoglycoside antibiotics, ethacrynic acid, high doses of salicylates, cisplatin, tubocurarine, succinylcholine, chloral hydrate, phenytoin, methotrexate, indomethacin, or lithium).
15. Administration of an investigational drug or implantation of investigational device, or participation in another interventional clinical trial, within 30 days prior to Screening.
16. Any surgical or medical condition which in the opinion of the investigator may interfere with participation in the study or which may affect the outcome of the study.
17. Positive urine drug screen at Screening or Baseline.
18. Blood alcohol concentration > 2 mg/dL (0.02%) at Screening.
19. Alcohol breath test > 2 mg/dL (0.02%) on admission to the CRU.
20. History of severe allergic or hypersensitivity reactions to furosemide or any component of the SCP-111 formulation (tromethamine or benzyl alcohol)

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
AUClast | 12 hours
  The area under the plasma concentration versus time curve from time 0 (pre-dose) to the last quantifiable time point.
AUCinf | 12 hours
  The area under the plasma concentration-time curve from time 0 (pre-dose) to time of last measurable plasma concentration.
Cmax | 12 hours
  Maximum observed plasma concentration of Furosemide
Tmax | 12 hours
  Time to achieve maximum observed Furosemide plasma concentration
λz | 12 hours
  Apparent plasma terminal-phase elimination rate constant
t½ | 12 hours
  Terminal-phase half life
V | 12 hours
  Systemic volume of distribution, terminal phase, for IV furosemide
Vz/F | 12 hours
  Apparent volume of distribution, terminal phase, for SC furosemide
CL | 12 hours
  Systemic clearance for IV furosemide
CL/F | 12 hours
  Apparent systemic clearance for SC furosemide
Urine Output | 6 hour, 8 hour and 12 hour
  Total Urine Output
Urinary Sodium | 6 hour, 8 hour and 12 hour
  Urinary sodium excretion
Urinary Potassium | 6 hour, 8 hour and 12 hour
  Urinary potassium excretion

SECONDARY OUTCOMES:
Adverse Events | Day 0 through Day 5 visit
  Adverse Events (AEs) and Serious Adverse Events (SAEs)
Injection Site Pain | 12 hours
  Injection site pain will be assessed using an 11-point scale where 0 is equivalent to no pain and 10 is equivalent to the worst possible pain. For IV administration, the 11-point pain scale will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Elixia EPCT, LLC, Tampa, Florida, United States